CLINICAL TRIAL: NCT07223957
Title: Using an Innovative Implementation Strategy to Increase the Translation of Effective Youth Violence Prevention Programs in Schools
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Injury Control Research Centers (ICRC) (Unknown)
Responsible Party: Principal Investigator, Belinda Hernandez, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-24-0976; RFA-CE-24-001 (Other Grant/Funding Number: Centers for Disease Control and Prevention); 5R49CE003712 (NIH)
Record Dates: First submitted 2025-10-30; First posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Bullying; Teen Dating Violence
MeSH Terms: conditions — Bullying

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iCHAMPS-YVP (Experimental)
  Interventions: Behavioral: iCHAMPS-YVP

INTERVENTIONS:
Behavioral: iCHAMPS-YVP — iCHAMPSS (CHoosing And Maintaining Effective Programs for Sex Education in Schools), a theory-based, online implementation strategy developed to increase the uptake of evidence-based sexual health programs (EBPs) in Texas schools. The intervention provides interactive tools, step-by-step guidance, and resources to assist school districts.

SUMMARY:
The purpose of this study is to Adapt the existing iCHAMPSS's tools to support school policies related to the adoption, implementation, and maintenance of effective youth bullying and dating violence prevention programs (iCHAMPS-YVP), to assess the usability (acceptability, ease of use, credibility, motivational appeal, and perceived helpfulness) of iCHAMPS-YVP in schools and to assess the feasibility of iCHAMPS-YVP with school staff to impact individual- (e.g.,knowledge, attitudes, and self-efficacy of school staff) and district-level (e.g., policy, readiness, and support) determinants of the adoption and implementation of effective youth violence prevention programs.

ELIGIBILITY:
Inclusion Criteria:

Hold one of the following positions:

* district or school administrator (e.g., health coordinators, instructional specialists, and curriculum coordinators)
* health and physical education teachers
* social and health service staff (e.g., nurses and counselors) in a Texas school district.

Exclusion Criteria:

* not holding a job in a Texas school district as a school stakeholder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Usability as assessed by the ease of use | Three weeks post iCHAMPS-YVP access
  This will be reported categorically on a Five-point Likert scale in the following categories from Very Easy, Kind of Easy, Kind of Hard, Very Hard, and Did Not Use
Change in Self-Efficacy as assessed by the iCHAMPS-YVP tasks | Baseline and 6 months post iCHAMPS-YVP access
  This will be reported categorically on a Four-point Likert scale in the following categories; not at all confident, somewhat confident, confident and very confident

SECONDARY OUTCOMES:
Current practices: dating violence prevention education | Baseline
  This will be reported categorically in the following categories;
  1. Yes, for middle school only
  2. Yes, for high school only
  3. Yes, for both middle and high school
  4. No, my district/school does not provide sexual health education to middle or high school
Current practices: bullying prevention education | Baseline
  This will be reported categorically in the following categories;
  1. Yes, for middle school only
  2. Yes, for high school only
  3. Yes, for both middle and high school
  4. No, my district/school does not provide sexual health education to middle or high school
Challenges that have prevented the district/school from implementing dating violence prevention education | Baseline
  This will be reported categorically in the following categories;
  1. There have been no challenges
  2. Lack of time to teach the curriculum
  3. No substitute teachers available
  4. Lack of curriculum resources (not including funding)
  5. Lack of funding
  6. Teacher comfort level with the content
  7. Lack of training opportunities for teachers
  8. Concerns about parents' reactions
  9. Concerns about students' reactions
  10. Concerns about reactions from administration or district
  11. Concerns about reactions from the community
  12. School or district policy regarding sexual health instruction
  13. Requirement of active parental consent
  14. Too many other district/school priorities
  15. Lack of Board of Trustees' approval of the curriculum
  16. Other (please specify):
Challenges that have been present when the district/school has implemented the curriculum for bullying prevention education instruction | Baseline
  This will be reported categorically in the following categories;
  1. There have been no challenges
  2. Lack of time to teach the curriculum
  3. No substitute teachers available
  4. Lack of curriculum resources (not including funding)
  5. Lack of funding
  6. Teacher comfort level with the content
  7. Lack of training opportunities for teachers
  8. Concerns about parents' reactions
  9. Concerns about students' reactions
  10. Concerns about reactions from administration or district
  11. Concerns about reactions from the community
  12. School or district policy regarding sexual health instruction
  13. Requirement of active parental consent
  14. Too many other district/school priorities
  15. Lack of Board of Trustees' approval of the curriculum
  16. Other (please specify):
Challenges to implementation that have prevented your district/school from adopting bullying prevention education | Baseline
  This will be reported categorically in the following categories;
  1. There have been no challenges
  2. Lack of time to teach the curriculum
  3. No substitute teachers available
  4. Lack of curriculum resources (not including funding)
  5. Lack of funding
  6. Teacher comfort level with the content
  7. Lack of training opportunities for teachers
  8. Concerns about parents' reactions
  9. Concerns about students' reactions
  10. Concerns about reactions from administration or district
  11. Concerns about reactions from the community
  12. School or district policy regarding sexual health instruction
  13. Requirement of active parental consent
  14. Too many other district/school priorities
  15. Lack of Board of Trustees' approval of the curriculum
  16. Other (please specify):
Intentions to replace current curriculum:dating violence prevention instruction | Baseline
  This will be reported categorically in the following categories;
  1. Yes
  2. No
  3. Don't know
Intentions to replace current curriculum: bullying prevention instruction | Baseline
  This will be reported categorically in the following categories;
  1. Yes
  2. No
  3. Don't know
Intentions to adopt an evidence-based program:dating violence prevention instruction | Baseline
  This will be reported categorically in the following categories;
  1. Yes
  2. No
  3. Don't know
Intentions to adopt an evidence-based program:bullying prevention instruction | Baseline
  This will be reported categorically in the following categories;
  1. Yes
  2. No
  3. Don't know
Acceptability | Three weeks post iCHAMPS-YVP access
  This will be reported categorically on a Five-point Likert scale in the following categories "Like a Lot", "Like a Little", "Dislike a Little", "Dislike a Lot", and "Did Not Use"
Helpfulness | Three weeks post iCHAMPS-YVP access
  This will be reported categorically on a three-point Likert scale in the following categories: "Less helpful", "As helpful", and "More helpful"
Perceived impact | Three weeks post iCHAMPS-YVP access
  This will be categorically reported in the following categories:
  1. yes
  2. no
  3. no opinion
Credibility | Three weeks post iCHAMPS-YVP access
  This will be categorically reported in the following categories:
  1. Accurate
  2. Inaccurate
  3. No opinion
Motivational Appeal | Three weeks post iCHAMPS-YVP access
  This will be categorically reported in the following categories:
  1. yes
  2. no
  3. no opinion
Change in Compatibility | Baseline and 6 months post iCHAMPS-YVP access
  this will be reported categorically on a Four-point Likert scale in the following categories: Strongly disagree disagree agree strongly agree
Change in Complexity | Baseline and 6 months post iCHAMPS-YVP access
  this will be reported categorically on a Four-point Likert scale in the following categories: Strongly disagree disagree agree strongly agree
Change in Perceived social systems support (for evidence-based programs) | Baseline and 6 months post iCHAMPS-YVP access
  this will be reported categorically on a Four-point Likert scale in the following categories: Not at all supportive supportive very supportive don't know
Change in Presence of organizational policy | Baseline and 6 months post iCHAMPS-YVP access
  This will be reported categorically in the following categories:
  1. No, and we have no plans to do so.
  2. No, but we are planning to implement an opt-in parental consent policy in the future.
  3. Yes, we are at an early stage of implementing an opt-in parental consent policy
  4. Yes, we have implemented an opt-in parental consent policy, but it is inconsistently implemented at the district or school.
  5. Yes, we have implemented an opt-in parental consent policy fully and systematically across the district or school.
  6. Don't know.
Challenges that have prevented your district/school from adopting dating violence prevention education | Baseline
  This will be reported categorically in the following categories:
  1. There have been no challenges
  2. Lack of time to teach the curriculum
  3. No substitute teachers available
  4. Lack of curriculum resources (not including funding)
  5. Lack of funding
  6. Teacher comfort level with the content
  7. Lack of training opportunities for teachers
  8. Concerns about parents' reactions
  9. Concerns about students' reactions
  10. Concerns about reactions from administration or district
  11. Concerns about reactions from the community
  12. School or district policy regarding sexual health instruction
  13. Requirement of active (i.e., "opt-in") parental consent
  14. Too many other district/school priorities
  15. Lack of Board of Trustees' approval of the curriculum
  16. Other (please specify):
Change in Intentions to use an evidence-based program | Baseline and 6 months post iCHAMPS-YVP access
  This will be reported categorically on a Six-point Likert in the following categories:
  Definitely will Probably will Probably will not Definitely will not Dont know not applicable
Change in Awareness/knowledge (of evidence-based programs) | Baseline and 6 months post iCHAMPS-YVP access
  This will be reported on a four point likert scale in the following categories:
  Strongly disagree disagree agree strongly agree
Change in Level of implementation | Baseline and 6 months post iCHAMPS-YVP access
  This will be reported categorically as follows:
  Prioritize: Refers to making violence prevention a priority for your district Assess: Refers to understanding your district's population, needs, and resources Select: Refers to identifying an evidence-based program that fits your district's population, needs, and resources Approve: Refers to getting your school board to approve an evidence-based program for use. Prepare: Refers to planning for complete and successful implementation of an approved evidence-based program Implement: Refers to implementing your evidence-based program with fidelity Maintain: Refers to improving and sustaining implementation of an evidence-based program over time.
Challenges that have been present when the district/school has implemented the curriculum for dating violence education instruction | Baseline
  This will be reported categorically in the following categories;
  1. There have been no challenges
  2. Lack of time to teach the curriculum
  3. No substitute teachers available
  4. Lack of curriculum resources (not including funding)
  5. Lack of funding
  6. Teacher comfort level with the content
  7. Lack of training opportunities for teachers
  8. Concerns about parents' reactions
  9. Concerns about students' reactions
  10. Concerns about reactions from administration or district
  11. Concerns about reactions from the community
  12. School or district policy regarding sexual health instruction
  13. Requirement of active parental consent
  14. Too many other district/school priorities
  15. Lack of Board of Trustees' approval of the curriculum
  16. Other (please specify):

CONTACTS AND LOCATIONS:
Overall Officials: Belinda Hernandez, PhD, MPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No